CLINICAL TRIAL: NCT01788982
Title: A Phase II Study Exploring the Safety and Efficacy of Nintedanib (BIBF1120) as Second Line Therapy for Patients With Either Differentiated or Medullary Thyroid Cancer Progressing After First Line Therapy.
Brief Title: Nintedanib(BIBF1120) in Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EORTC-1209; 2012-004295-19 (EudraCT Number)
Record Dates: First submitted 2013-02-08; First posted 2013-02-11 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Medullary Thyroid Cancer (MTC); Differentiated Thyroid Cancer (DTC)
Keywords: Thyroid Cancer; Medullary thyroid cancer (MTC); Differentiated thyroid cancer (DTC)
MeSH Terms: conditions — Carcinoma, Medullary; Thyroid Neoplasms | interventions — nintedanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nintedanib (Experimental): Nintedanib should be administered orally at a dose of 200 mg twice daily.
  Interventions: Drug: Nintedanib
- Placebo (Placebo Comparator): Placebo should be administered orally at a dose of 200 mg twice daily. Cross-over to nintedanib is allowed after progression.
  Interventions: Drug: Nintedanib; Drug: Placebo

INTERVENTIONS:
Drug: Nintedanib — Nintedanib should be administered orally at a dose of 200 mg twice daily.
  Other Names: BIBF1120
Drug: Placebo
  Arms: Placebo

SUMMARY:
For the treatment of thyroid cancer with the so called targeted therapy the angiogenesis pathway has several potential targets. The Receptors for Vascular endothelial growth factor (VEGF) and especially VEGFR-2 is considered to be crucial for the initiation of the formation as well as the maintenance of tumor vasculature.

In thyroid cancer these VEGF receptors (VEGFR-1, VEGFR-2), VEGF itself and receptors of the fibroblast growth factor (FGF) and for the platelet-derived growth factor (PDGF) are often overexpressed. Other cells as pericytes and smooth muscle cells that are also involved in tumor angiogenesis express these receptors as well.

Inhibitors of the VEGFR or PDGFR pathway have been tested in thyroid cancer with positive results. However there is no treatment that is generally considered as standard of care for patients with differentiated thyroid cancer (DTC) or medullar thyroid cancer (MTC) who have progressed on one line of therapy. The classical cytotoxic chemotherapy has not shown a clinically meaningful benefit yet.

Nintedanib is a triple angiogenesis inhibitor which inhibits receptors of VEGF, FGF and PDGF. Therefore it might act not only on endothelial cells but also on pericytes and smooth muscle cells. Nintedanib also interacts with other kinases such as RET. Because of this multi-kinase activity rationale exists to investigate the effect in MTC and DTC.

Because it targets these three major angiogenesis signaling pathways it might prevent further tumor growth and related tumor escape mechanisms. Therefore nintedanib may be active in patients who have progressed on agents that target only one pathway.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed differentiated or medullary thyroid cancer by local pathologist.
* Available tumor tissue at the time of initial diagnosis for histology review. The provision of tumor tissue for histology review is mandatory for every patient/site.
* Locally advanced or metastatic disease deemed incurable by surgery, radiotherapy and/or radioactive iodine (RAI).
* No current symptomatic brain metastases or if previously present, must have been treated at least two months before randomization. CT or MRI scan of the brain is mandatory (within 4 weeks prior to randomization) to assess the presence or not of brain metastases.
* Patients must have measurable lesion with documented progression during the 12 months prior to randomization, according to RECIST V.1.1. Patients who were withdrawn from first line treatment due to toxicity without documented disease progression or who received placebo (in the context of a clinical trial) as prior treatment are not eligible.
* Patients must have received one or 2 prior line of treatment (but no more than two) and must be off treatment for at least 4 weeks prior to randomization.
* Age ≥18 years.
* Performance status (PS) 0-1 (WHO, Appendix C).
* Life expectancy of more than 12 weeks.
* No history of other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix or basal cell or spinocellular carcinoma of the skin.
* No ongoing treatment related toxicity due to prior treatment > grade I (except alopecia).
* Adequate organ function, evidenced by the following laboratory results within 3 weeks prior to randomization: (patients with a buffer range from the normal values of +/- 5% for hematology and +/- 10% for biochemistry [with the EXCEPTION of Glomerular Filtration Rate] are acceptable)

  * Absolute neutrophil count > 1500 cells/mm3
  * Platelet count > 100,000 cells/mm3
  * Hemoglobin > 8.5 g/dL
  * Total bilirubin within normal limits
  * SGOT (AST), SGPT (ALT), and alkaline phosphatase ≤ 1.5× ULN (or ≤ 2.5× ULN) in the case of presence of liver metastases)
  * Glomerular Filtration Rate (GFR) ≥ 45 ml/min according to Cockcroft and Gault Formula (see Appendix E.).
  * Proteinuria CTC-AE < 2
  * Coagulation parameters: International normalized ratio (INR) ≤ 2, prothrombin time (PT) and partial thromboplastin time (PTT) ≤ 1.5x institutional ULN
* No history of significant cardiac disease defined as:

  * Symptomatic CHF (NYHA classes III-IV, see Appendix D)
  * High-risk uncontrolled arrhythmias, i.e. atrial tachycardia with a heart rate > 100/min at rest, significant ventricular arrhythmia (ventricular tachycardia) or higher-grade AV-block (second degree AV-block Type 2 [Mobitz 2] or third degree AV-block)
  * No prolongation of corrected QT interval (QTc) > 480 msecs,
  * History of myocardial infarction within 12 months prior to randomization
  * Clinically significant valvular heart disease
  * No angina pectoris requiring anti-angina treatment
* No current uncontrolled hypertension (persistent systolic > 180 mmHg and/or diastolic > 100 mmHg) (with or without medication). Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry.
* No evidence of active bleeding or bleeding diathesis.
* No cerebrovascular accident at any time in the past, transient ischemic attack, deep venous thrombosis (DVT) or pulmonary embolism in the past 6 months.
* Therapeutic anticoagulation (except low-dose heparin and/or heparin flush as needed for maintenance of an in-dwelling intravenous devise) or anti-platelet therapy (except for low-dose therapy with acetylsalicylic acid < 325mg per day) is not allowed.
* No history of clinically significant gastrointestinal disorders including: malabsorption syndrome, major resection of the stomach or small bowel that could affect the absorption of study drug, active peptic ulcer disease, known intraluminal metastatic lesions with risk of bleeding, inflammatory bowel disease, ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation. No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment.
* No current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease; wound healing disorders; ulcers; or bone fractures, known infection with HIV, active hepatitis B and/or hepatitis C virus) or any other systemic disease/symptoms that may hamper compliance to study protocol, according to physician's judgment.
* No major surgical procedure or significant traumatic injury within 28 days prior to randomization or anticipation of the need for major surgery during the course of study treatment and/or presence of any non-healing wound, fracture, or ulcer.
* No history of receiving any investigational treatment within 28 days prior to randomization.
* Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test within 72 hours prior to the first dose of study treatment.
* Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 6 months after the last study treatment. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 6 months after the last study treatment.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

  * Tissue availability for central confirmation of the histological diagnosis is mandatory. All other TR projects are optional for the patient and a separate consent form for these will be provided to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-05; Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 2,5 years from FPI
  This study will use RECIST 1.1 to measure PFS

SECONDARY OUTCOMES:
Occurence of Adverse Events | 2,5 years from FPI
  This study will use the International Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, for adverse event reporting.
Response Rate | 2,5 years from FPI
  This study will use RECIST 1.1 to measure RR
Duration of response | 2,5 years form FPI
  This study will use RECIST 1.1 to measure duration of response
Exploration of the molecular mechanisms of action of drug | 3 years from FPI
  The biomarker study in this protocol is exploratory in nature.Spearman Correlation Coefficient will be computed to quantify the relationship between biomarkers and between biomarkers and clinical parameters (e.g. age). Fisher's exact test or Wilcoxon rank sum test will be used to assess the significance of these relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schlumberger, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (27):
- Belgium (6):
  - A.Z. St. Jan, Bruges
  - Hopitaux Universitaires Bordet-Erasme - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem, Antwerpen
  - Universitair Ziekenhuis Gent, Ghent
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
- Odense University Hospital, Odense, Denmark
- France (9):
  - CHU d'Angers, Angers
  - Institut Bergonie, Bordeaux
  - Centre Regional Francois Baclesse, Caen
  - Centre Georges-Francois-Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Assitance Publique - Hopitaux de Paris - Hopital Saint-Louis, Paris
  - Assistance Publique - Hopitaux de Paris - La Pitié Salpétrière, Paris
  - Centre Jean Godinot, Reims
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Ludwig-Maximilians-Universitaet Muenchen - Klinikum der Universitaet Muenchen - Campus Grosshadern, Munich
  - Universitaetsklinikum Wuerzburg, Würzburg
- Italy (2):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
- Netherlands (3):
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Centre, Leiden
  - Radboud University Medical Center Nijmegen, Nijmegen
- Maria Sklodowska-Curie Memorial Cancer Centre, Warsaw, Poland
- Hospital General Vall D'Hebron, Barcelona, Spain
- United Kingdom (2):
  - Royal Marsden Hospital - Sutton, Surrey, Sutton, Surrey
  - NHS Greater Glasgow and Clyde - Beatson West of Scotland Cancer Centre - Gartnavel General Hospital, Glasgow